CLINICAL TRIAL: NCT05792098
Title: Percutaneous Dilatational Tracheostomy and Thyroid Isthmus Penetration
Acronym: PETRIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Military University Hospital, Prague (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PETRIS_01
Record Dates: First submitted 2023-03-07; First posted 2023-03-30 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Tracheostomy Complication
Keywords: percutaneous dilatational tracheostomy; ultrasound; mechanical ventilation
MeSH Terms: interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard procedure group (Active Comparator): The standard procedure group will undergo PDTS by the attending physician in the standard manner based on clinical examination and anatomical landmarks using bronchoscopic control.
  Interventions: Procedure: percutaneous dilatational tracheostomy (PDTS); Diagnostic Test: Bronchoscopy
- Ultrasound navigated group (Active Comparator): Ultrasound navigated group, the attending physician will additionally use ultrasound navigation during the procedure.
  Interventions: Procedure: percutaneous dilatational tracheostomy (PDTS); Diagnostic Test: Ultrasound examination; Diagnostic Test: Bronchoscopy

INTERVENTIONS:
Procedure: percutaneous dilatational tracheostomy (PDTS) — Tracheostomy made by percutaneous dilatational technique
Diagnostic Test: Ultrasound examination — Ultrasound verification of guidewire position
  Arms: Ultrasound navigated group
Diagnostic Test: Bronchoscopy — Bronchoscopic control of guidewire position

SUMMARY:
A prospective randomized interventional study will be conducted in the Military University Hospital Prague at the department of Anesthesiology and Intensive care. The incidence of thyroid isthmus penetration will be evaluated during percutaneous dilatational tracheostomy in two groups (ultrasound-guided puncture vs. standard approach using only anatomical landmarks).

DETAILED DESCRIPTION:
A prospective randomized interventional study will be conducted in the Military University Hospital Prague at the department of Anesthesiology and Intensive care. Patients indicated by the attending physician to percutaneous dilatational tracheostomy (PDTS) due to long-term need for mechanical ventilation will be randomly divided into two groups. The standard procedure group will undergo PDTS by the attending physician in the standard manner based on clinical examination and anatomical landmarks using bronchoscopic navigation. In the second group, the attending physician will additionally use ultrasound navigation during the procedure. After insertion of the guidewire, before dilation is performed, patients in both groups will be examined by ultrasound by an independent physician - the study investigator - who will verify the position of the guidewire and its relationship to the surrounding structures. In case of malposition of the guidewire (unacceptable lateral or craniocaudal), the penetration site will be adjusted and the PDTS completed.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years and older
* long-term need for mechanical ventilation

Exclusion Criteria:

* not willing to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
The guidewire penetration through the thyroid isthmus. | During procedure
  Incidence of guidewire penetration through the thyroid isthmus in standard and ultrasound navigated percutaneous dilatational tracheostomy.
Monitoring the incidence of early postoperative complications. | Up to 10 days
  The incidence of bleeding from tracheostomy canal during hospitalization depending on guidewire position, defined as the need for any intervention to stop the bleeding.
  The incidence of tracheostomy canal infection during hospitalization depending on guidewire position, defined as the presence of any clinical signs of inflammation (swelling, redness, pain, secretion production, dehiscence).

SECONDARY OUTCOMES:
Using ultrasound examination as a tool for PDTS navigation in terms of correct puncture site. | During procedure
  Monitoring the frequency of guidewire position changes based on ultrasound examination.

OTHER OUTCOMES:
Ultrasound-based contraindication rate of percutaneous dilatational tracheostomy. | During procedure
  Monitoring the incidence of tracheostomy technique change from planned percutaneous dilatation to surgical approach based on ultrasound examination.

CONTACTS AND LOCATIONS:
Overall Officials: Ilona Trtíková, Mgr., Ph.D., Study Chair — CHARLES UNIVERSITY, FIRST FACULTY OF MEDICINE AND GENERAL UNIVERSITY HOSPITAL IN PRAGUE
Locations (1):
- Military University Hospital Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gobatto ALN, Besen BAMP, Tierno PFGMM, Mendes PV, Cadamuro F, Joelsons D, Melro L, Carmona MJC, Santori G, Pelosi P, Park M, Malbouisson LMS. Ultrasound-guided percutaneous dilational tracheostomy versus bronchoscopy-guided percutaneous dilational tracheostomy in critically ill patients (TRACHUS): a randomized noninferiority controlled trial. Intensive Care Med. 2016 Mar;42(3):342-351. doi: 10.1007/s00134-016-4218-6. Epub 2016 Feb 1. PMID 26831676
- [Background] Plata P, Gaszynski T. Ultrasound-guided percutaneous tracheostomy. Anaesthesiol Intensive Ther. 2019;51(2):126-132. doi: 10.5114/ait.2019.86277. PMID 31268274